CLINICAL TRIAL: NCT00005809
Title: Computerized Tomographic Colonography: Performance Evaluation in a Multicenter Setting
Brief Title: Computerized Tomographic Colonography Compared With Standard Diagnostic Procedures in Detecting Colorectal Neoplasia
Acronym: ACRIN 6656
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000067802; ACRIN-6656; CA80098 (Other Grant/Funding Number: NCI CIP)
Record Dates: First submitted 2000-06-02; First posted 2004-04-19 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: computed tomography
Procedure: diagnostic colonoscopy

SUMMARY:
RATIONALE: New diagnostic procedures such as computed tomographic colonography may provide a less invasive method of identifying patients who have colorectal neoplasia.

PURPOSE: Diagnostic study to compare the effectiveness of computerized tomographic colonography with that of standard diagnostic procedures in detecting colorectal neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare retrospectively the accuracy of computerized tomographic colonography (CTC) vs pathology and colonoscopy in the detection of clinically important colorectal neoplasia, defined as at least one proven lesion with a diameter measuring at least 1 cm. II. Compare the physician image display preferences and interpretation time across three viewing platforms for CTC images.

OUTLINE: This is a retrospective, multicenter study. Radiologists evaluate each patient's optimal diagnostic computerized tomographic colonography (CTC) data. Patients' CTC findings are evaluated by a radiologist at a central facility using an imaging display software platform from General Electric, Vital Images, or the Mayo Clinic. CTC findings are compared with conventional colonoscopy findings and pathologic analysis. A comparison is made between physician image display preferences and interpretation time across three viewing platforms for CTC images.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: The following case material must be submitted for each patient: No colonic diseases except polyps, cancer, or diverticulosis Optimal diagnostic computerized tomographic colonography (CTC) data with computed tomography acquisition parameters that meet the following minimal standards: Slice thickness no greater than 5 mm Reconstruction interval no greater than 3 mm Pitch no greater than 2 Anatomic coverage of the entire colorectum Supine and prone data sets Complete colonoscopy performed within 30 days following CTC by a board certified gastroenterologist or a physician with at least 3 years of colonoscopic experience Pathology reports for all endoscopically or surgically removed colorectal lesions with the exception of polyps that are inadvertently dropped at the time of retrieval Photograph or videotape record of dropped lesion allowed as proof of its existence All studies are allowed including those with lesions less than 1 cm, lesions at least 1 cm, or no lesions Report documents size, site, stage, grade, and type of colorectal cancers; size, site, degree of dysplasia, and type of colorectal adenomas; and types of other lesions (e.g., inflammatory, vascular, ulcerative) Demographic data including patient's age, sex, ethnic background, symptoms, risk factors, and relevant clinical history

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2000-10 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Daniel Johnson, MD, Study Chair — Mayo Clinic
Locations (11):
- United States (11):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Result] Johnson CD, Toledano AY, Herman BA, Dachman AH, McFarland EG, Barish MA, Brink JA, Ernst RD, Fletcher JG, Halvorsen RA Jr, Hara AK, Hopper KD, Koehler RE, Lu DS, Macari M, Maccarty RL, Miller FH, Morrin M, Paulson EK, Yee J, Zalis M; American College of Radiology Imaging Network A6656. Computerized tomographic colonography: performance evaluation in a retrospective multicenter setting. Gastroenterology. 2003 Sep;125(3):688-95. doi: 10.1016/s0016-5085(03)01058-8. PMID 12949715